CLINICAL TRIAL: NCT03040804
Title: A Phase I Study of Low Dose Radiotherapy for Advanced Hidradenitis Suppurativa
Brief Title: Low Dose Radiotherapy for Advanced Hidradenitis Suppurativa
Acronym: RTHS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Infeasibility to continue study.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Steven R Cohen, Chief of Dermatology at Montefiore, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-7228
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Hidradenitis Suppurativa; Hidradenitis
Keywords: hidradenitis suppurativa; HS; radiotherapy
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis | interventions — Radiotherapy; Brachytherapy

STUDY DESIGN:
Intervention Model Description: Simon two-stage design. In the first stage, 6 patients will be enrolled. If the patients in the study do not meet the termination criteria then the study will extend to a second stage and a maximum of 20 patients will be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low Dose Radiotherapy (Experimental): Patients will receive skin-directed radiotherapy, using a total prescription dose of 7.5 gy in five fractions of 1.5 gy over one week
  Interventions: Radiation: Low dose Radiotherapy

INTERVENTIONS:
Radiation: Low dose Radiotherapy — Subjects in this protocol will only receive radiotherapy directed at one region, typically the region that is most bothersome to the patient. Patients will receive a total radiotherapy dose 7.5 Gy in five daily fractions of 1.5 Gy.
  Other Names: Brachytherapy

SUMMARY:
To establish the safety of radiotherapy in the treatment of advanced hidradenitis suppurativa. Patients will receive radiotherapy treatment over one week and then they will be followed for the next three months.

DETAILED DESCRIPTION:
This is a phase I clinical trial using a Simon-two stage design to establish the safety of radiotherapy in the treatment of advanced hidradenitis suppurativa (HS). In the first six months, 6 patients will be enrolled, if the patients in the study do not meet the termination criteria, then the study will extend to a second stage. A maximum of 20 patients will be enrolled. Patients will be treated with skin-directed radiotherapy, using a total prescription dose of 7.5 Gy in five fractions of 1.5 Gy over one week. Patients will then be seen in the HS specialty clinic at Montefiore Medial Center for at least three months. Quality of life changes, immunohistochemical changes, and cutaneous discharge will also be evaluated during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hidradenitis Suppurativa made at the Montefiore Hidradenitis Suppurativa Treatment Center, with Hurley Stage 2-3 (defined as recurrent abscesses or boils with diffuse or broad involvement, multiple interconnected sinus tracts in the whole area)
* Failed maximal medical therapy for Hidradenitis Suppurativa or ineligible for "standard" medical therapy or surgery
* Age > 20 years
* Women of childbearing age: must have a negative pregnancy test within 72 hours prior to the start of study therapy and agree to an adequate method of contraception throughout treatment and for at least 4 weeks after study contraception.

Exclusion Criteria:

* Pregnant women
* Individuals < 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Cohen, MD, MPH, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Montefiore Hidradenitis Suppurativa Multispecialty clinic — http://www.montefiore.org/hidradenitis-suppurativa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Radiotherapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Dose Radiotherapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 70 [67 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1
  Caucasian | 1
Region of Enrollment [Number; unit: participants]
  United States | 2
Improvement in hidradenitis suppurativa lesion size [Number; unit: participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HS Who Experience Treatment-related Grade ≥3 Adverse Events During Radiotherapy or Within 3 Months of Radiotherapy Completion, Assessed Using CTCAE Version 4.0
Description: Number of participants with HS who experience treatment-related CTCAE version 4.0 Grade ≥3 adverse events during radiotherapy or within 3 months of radiotherapy completion. Common Terminology Criteria for Adverse Events (CTCAE) is an internationally accepted standard for defining and categorizing adverse events based on severity of reported adverse events. The grading scheme is from 1 (least severe) to 5 (most severe). For radiotherapy associated adverse events, CTCAE version 4.0 will be applied to "Rash: dermatitis associated with radiation".
  Grade 1. Mild: Faint erythema or dry desquamation. Grade 2. Moderate: Moderate to brisk erythema; patchy moist desquamation, mostly confined to skin folds and creases; moderate edema.
  Grade 3. Severe: Moist desquamation other than skin folds and creases; bleeding induced by minor trauma or abrasion.
  Grade 4. Life threatening: Skin necrosis or ulceration of full thickness dermis; spontaneous bleeding from involved site.
  Grade 5
Time Frame: follow up for 3-6 months post treatment
Population: Patients with Hidradenitis Suppurativa (HS) Hurley Stage 2-3.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Radiotherapy
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Changes in NIH Patient-Reported Outcomes Measurement Information System (PROMIS).
Description: Evaluation of the efficacy of radiotherapy in improvement of patient's quality of life using patient reported outcome measures, including pain interference and physical functioning at 3 months (and optionally at 6 months and 12 months) after treatment.
Time Frame: 6 months - 1 year post treatment
Population: Due to COVID-19 pandemic, patient safety was prioritized and the study was terminated early. Participant outcome measures were not performed.
Arm/Group | Low Dose Radiotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Evaluation of Radiotherapy Associated Hidradenitis Suppurativa Lesions.
Description: Hematoxylin and Eosin (H&E) stain and immunohistochemistry stains will be performed on skin biopsy specimens to investigate histological changes following radiotherapy for advanced hidradenitis suppurativa lesions.
Time Frame: 3-6 months post treatment
Population: Due to COVID-19 pandemic, patient safety was prioritized and the study was terminated early. Participant outcome measures were not completed.
Arm/Group | Low Dose Radiotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Two participants were observed in relation to baseline radiotherapy treatment for an average of 6 months.
Groups:
- Low Dose Radiotherapy: Patients will receive skin-directed radiotherapy, using a total prescription dose of 7.5 gy in five fractions of 1.5 gy over one week
  Low dose Radiotherapy: Subjects in this protocol will only receive radiotherapy directed at one region, typically the region that is most bothersome to the patient. Patients will receive a total radiotherapy dose 7.5 Gy in five daily fractions of 1.5 Gy.
  No adverse event reported to date.
Arm/Group | Low Dose Radiotherapy
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT03040804/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT03040804/ICF_001.pdf